CLINICAL TRIAL: NCT01672359
Title: The Effect of Whole-Food Dietary Supplementation on Cognitive and Immune Functioning and Quality of Life in Healthy Older Adults
Brief Title: Evaluating Whole Foods Supplementation on Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Standard Process Inc. (Industry)
Responsible Party: Principal Investigator, John E. Lewis, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20090985
Record Dates: First submitted 2012-08-20; First posted 2012-08-24 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Sub-optimal Cognitive Function; Sub-optimal Immune Function
Keywords: cognitive functioning; immune function; cytokines; growth factors; quality of life; dietary supplementation; Ginkgo biloba; Improvement of cognitive function
MeSH Terms: interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ginkgo Synergy® and Choline (Experimental): Ginkgo Synergy® (120 mg/day Ginkgo biloba leaf with 80 mg/day Ginkgo biloba whole extract combined with 40 mg/day Grape Seed extract) and Choline (700 mg choline/day)
  Interventions: Dietary Supplement: Ginkgo Synergy® and Choline
- OPC Synergy® and Catalyn (Experimental): OPC Synergy® (100 mg/day of Grape Seed extract with 50 mg/day Green Tea extract (60% catechins)) and Catalyn® (1,248 IU/day of Vitamin D, 4,800 IU/day of Vitamin A, combined with vitamin C, thiamine, riboflavin, and vitamin B6)
  Interventions: Dietary Supplement: OPC Synergy® and Catalyn
- Placebo (Placebo Comparator): cellulose pills to simulate actual products
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ginkgo Synergy® and Choline — 3 tablets 2 times per day with breakfast and dinner over 6 months
  Arms: Ginkgo Synergy® and Choline
Dietary Supplement: OPC Synergy® and Catalyn — 3 tablets 2 times per day with breakfast and dinner over 6 months
  Arms: OPC Synergy® and Catalyn
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
A six-month study which investigated the effect of Ginkgo Synergy® and Choline or OPC Synergy® and Catalyn® on cognitive and immune function markers and quality of life among healthy older adults with no history of significant cognitive deficits

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age and older
* English speaking
* Not living in a skilled or intermediate care level nursing facility
* No use of dietary supplements for cognitive functioning two weeks before enrolling in the study and during the length of the trial
* A Mini-Mental State Exam (MMSE) score ≥ 23

Exclusion Criteria:

* A cognitive deficit greater than that indicated according to the MMSE score
* A clinical diagnosis of AD and/or related disorders
* A psychiatric diagnosis of schizophrenia, other psychotic disorders, bipolar disorder, major depression with psychotic features, delirium, and alcohol or substance abuse/dependence
* Bleeding disorders
* Aphasia or sensory, motor, and/or visual disturbances that would have interfered with psychometric tests
* Gastrointestinal disorders causing impaired absorption of the study supplements
* Insulin-dependent diabetes
* Major conditions such as cardiovascular, pulmonary, renal, thyroid, hepatic, gastrointestinal, or seizure
* Hematologic or oncologic disorders treated with chemotherapy in the previous two years
* Active chemotherapy or radiation treatment for cancer
* Current cigarette smoking
* More than three major medical or psychiatric hospitalizations in the past year
* Diagnosis of a terminal illness
* A T score > 70 on the Global Severity Index of the Brief Symptoms Inventory (BSI)
* A score ≥ 29 on the Beck Depression Inventory-II (BDI) (15)
* Prescription and OTC sympathomimetic amines and antihistamines within 2 days of an assessment visit
* Cognition enhancing drugs consumption such as Donepezil, Rivastigmine, Galantamine, and Tacrine
* Coumadin, tricyclic antidepressants, antipsychotics, and anticonvulsants
* Cognition-enhancing supplements, herbs, or antioxidants that could not be stopped during the trial
* Participating in a concurrent trial for drugs, supplements, or treatment that affects behavior or cognitive function

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Cognitive Measures | 6 months
  The measures included the MMSE, the Stroop Color and Word Test (SCWT), the Trail Making Test Parts A and B (TMT-A, TMT-B), the Controlled Oral Word Association test (COWA), the Digit Symbol subtest of the Wechsler Adult Intelligence Scale, Third Edition (WAIS-III), and the Hopkins Verbal Learning Test-Revised (HVLT-R)

SECONDARY OUTCOMES:
Quality of Life Measures | 6 months
  Quality of Well-Being Scale (QWBS) Medical Outcomes Study Short Form 36 (SF 36) Beck Depression Inventory (BDI) Beck Anxiety Inventory (BAI)
Immune Function Markers | 6 months
  interleukin [IL]-2, IL-4, IL-6, IL-8, IL-10, IL-1α, IL-1β, interferon [IFN]-γ, tumor necrosis factor [TNF]-α, monocyte chemotactic protein [MCP]-1, vascular endothelial growth factor [VEGF], and epidermal growth factor [EGF]

CONTACTS AND LOCATIONS:
Overall Officials: John Lewis, PhD, Principal Investigator — University of Miami
Locations (1):
- Clinical Research Building, Miami, Florida, United States

REFERENCES:
- [Derived] Lewis JE, Melillo AB, Tiozzo E, Chen L, Leonard S, Howell M, Diaz J, Gonzalez K, Woolger JM, Konefal J, Paterson E, Barnes D. A double-blind, randomized clinical trial of dietary supplementation on cognitive and immune functioning in healthy older adults. BMC Complement Altern Med. 2014 Feb 4;14:43. doi: 10.1186/1472-6882-14-43. PMID 24495355